CLINICAL TRIAL: NCT03318341
Title: TheraBracelet Phase I Small Business Technology Transfer Research (STTR) - The 1st and Only Wearable to Instantly Improve Hand Function
Brief Title: TheraBracelet Phase I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TheraBracelet, Inc. (Industry)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R41HD090792-01A1 (NIH)
Record Dates: First submitted 2017-09-20; First posted 2017-10-23 (Actual); Results first posted 2019-03-06 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Hand Function; Stroke; Upper Extremity; Hemiparesis; Cerebrovascular Accident; Stroke Rehabilitation
Keywords: physical stimulation; Subliminal stimulation; stroke rehabilitation; upper extremity; paresis; patient safety
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: The study will use a 2×2 crossover design. Participants will be randomly assigned to either the treatment or control condition for the first month, followed by a 2-week washout period and then crossover to the other condition.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be blinded to the conditions, since they will not perceive any vibration for both conditions. The researcher conducting the evaluations with participants will also be blinded with the following procedure: A person outside the university will generate a random condition assignment sequence and send a custom program to the researcher to use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Real then Sham (Other): Participants are instructed to wear the TheraBracelet device on the affected wrist every day for at least 8 hours/day during their daily activity for 1 month. After 2-week washout, participants are again instructed to wear the device on the affected wrist every day for at least 8 hours/day during their daily activity for 1 month. The device applies real stimulation in the first month. The device applies sham stimulation in the second month. The stimulation is imperceptible. Thus, participants do not perceive stimulation in either month.
  Interventions: Device: Real Stimulation; Device: Sham Stimulation
- Sham then Real (Other): Participants are instructed to wear the TheraBracelet device on the affected wrist every day for at least 8 hours/day during their daily activity for 1 month. After 2-week washout, participants are again instructed to wear the device on the affected wrist every day for at least 8 hours/day during their daily activity for 1 month. The device applies sham stimulation in the first month. The device applies real stimulation in the second month. The stimulation is imperceptible. Thus, participants do not perceive stimulation in either month.
  Interventions: Device: Real Stimulation; Device: Sham Stimulation

INTERVENTIONS:
Device: Real Stimulation — The device applies wrist vibration at a subthreshold (imperceptible) level.
Device: Sham Stimulation — The device applies no vibration.

SUMMARY:
This project aims to test a new technology that may improve hand function impaired from a stroke, thereby improving independence and quality of life.

DETAILED DESCRIPTION:
Post-stroke hand impairment is highly prevalent and severely restricts functional ability and independence. Yet, there is no assistive device to help hand function at home, every day, during activities of daily living. Existing devices such as hand-opening orthoses are expensive, uncomfortable, bulky, and meant for use during short therapy sessions as opposed to during daily living. Thus their impact is limited. Consequently, the development of efficacious and affordable assistive device is of importance. This project addresses this critical gap by providing an innovative patent-pending technology. The "TheraBracelet" is a wristband applying imperceptible vibration to skin. TheraBracelet is efficacious, as it has been shown to immediately improve chronic stroke survivors' touch sensation and hand dexterity in previous studies. TheraBracelet is affordable by using only a low-cost vibrator. TheraBracelet is also translational, because a vibrator strategically placed at the wrist does not interfere with dexterous finger motions, and it is low-risk by involving only imperceptible vibration on skin. These practicalities assure easy adoption in home environment for large impact on sensorimotor impairment. The essential next step, thus the objective of this Phase I project, is to determine the feasibility and safety of using this assistive device all day every day for a month during daily activity. This objective will be accomplished in a double-blinded, randomized, controlled, crossover design study. Feasibility (compliance of using the device everyday) and safety will be assessed for the real vibration condition compared to the sham vibration condition (wearing the device without vibration). The feasibility and safety level comparable to those of wearing a watch and of a comparable FDA-approved device will support viability of TheraBracelet with necessary regulatory approvals. This project is expected to lead to an assistive wristband that increases hand function during activities of daily living for a large number of stroke survivors with hand impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Time since stroke: > 3 months
* Those with at least some movement in the affected upper limb
* Ability to put on the device at home
* Ability to perform the Box and Block Test with a score > 0

Exclusion Criteria:

* Comorbidity such as neuropathy, orthopaedic conditions in the hand
* Compromised skin integrity of the hand/wrist.
* Participation in an upper limb rehabilitation program concurrently
* Pregnancy
* A language barrier or cognitive impairment that precludes following
* Individuals whose swelling changes dramatically during the day
* Participant has received Botulinum toxin injection in the past 3 months
* Inability or unwillingness of subject or legal guardian/representative to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Na Jin Seo, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request.
Time Frame: The data will become available within 1 year from the study completion date for 6 years.
Access Criteria: De-identified data only

REFERENCES:
- [Derived] Seo NJ, Enders LR, Fortune A, Cain S, Vatinno AA, Schuster E, Ramakrishnan V, Feng W. Phase I Safety Trial: Extended Daily Peripheral Sensory Stimulation Using a Wrist-Worn Vibrator in Stroke Survivors. Transl Stroke Res. 2020 Apr;11(2):204-213. doi: 10.1007/s12975-019-00724-9. Epub 2019 Aug 23. PMID 31444692

RESULTS

PARTICIPANT FLOW:
Groups:
- Real Then Sham: Participants are instructed to wear the TheraBracelet device on the affected wrist every day for at least 8 hours/day during their daily activity for 1 month. After 2-week washout, participants are again instructed to wear the device on the affected wrist every day for at least 8 hours/day during their daily activity for 1 month. The device applies real stimulation in the first month. The device applies no stimulation in the second month. The stimulation is imperceptible. Thus, participants do not perceive stimulation in either month.
  Real Stimulation: The device applies wrist vibration at a subthreshold (imperceptible) level.
  Sham Stimulation: The device applies no vibration.
- Sham Then Real: Participants are instructed to wear the TheraBracelet device on the affected wrist every day for at least 8 hours/day during their daily activity for 1 month. After 2-week washout, participants are again instructed to wear the device on the affected wrist every day for at least 8 hours/day during their daily activity for 1 month. The device applies no stimulation in the first month. The device applies real stimulation in the second month. The stimulation is imperceptible. Thus, participants do not perceive stimulation in either month.
  Real Stimulation: The device applies wrist vibration at a subthreshold (imperceptible) level.
  Sham Stimulation: The device applies no vibration.
Period: Month 1
Arm/Group | Real Then Sham | Sham Then Real
Started | 13 | 13
Completed | 13 | 12
Not Completed | 0 | 1
Period: Month 2
Arm/Group | Real Then Sham | Sham Then Real
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real Then Sham | Sham Then Real | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11) | 58 (10) | 60 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Safety - Occurrence of Device-Related Adverse Events (AE)
Description: Any worsening of hand sensation, dexterity, grip strength, upper limb pain, swelling, spasticity, skin irritation, or any other adverse events (assessed every week) that sustained until the end of the month or occurred at the end of the month.
Time Frame: Two 1-month durations
Measure: Count of Participants; unit: Participants
Groups:
- Real Then Sham: Receive real stimulation for 1 month, then sham stimulation for 1 month.
- Sham Then Real: Receive sham stimulation for 1 month, then real stimulation for 1 month.
Arm/Group | Real Then Sham | Sham Then Real
Number analyzed (Participants) | 13 | 12
Participants
  AE Month 1 | 2 | 4
  AE Month 2 | 0 | 1

2. Primary Outcome: Feasibility - User Compliance in Wearing the Device
Time Frame: Two 1-month durations
Measure: Count of Participants; unit: Participants
Arm/Group | Real Then Sham | Sham Then Real
Number analyzed (Participants) | 13 | 12
Participants
  Compliance Month 1 | 13 | 12
  Compliance Month 2 | 13 | 12

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 2.5 month study period.
Groups:
- Real Then Sham - Month 1 (Real): Receive real stimulation for month 1
- Sham Then Real - Month 1 (Sham): Receive sham stimulation for month 1
- Real Then Sham - Month 2 (Sham): Receive sham stimulation for month 2.
- Sham Then Real - Month 2 (Real): Receive real stimulation month 2.
Arm/Group | Real Then Sham - Month 1 (Real) | Sham Then Real - Month 1 (Sham) | Real Then Sham - Month 2 (Sham) | Sham Then Real - Month 2 (Real)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/13 | 2/12 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 8/13 | 6/12 | 6/13 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real Then Sham - Month 1 (Real) (N=13) | Sham Then Real - Month 1 (Sham) (N=12) | Real Then Sham - Month 2 (Sham) (N=13) | Sham Then Real - Month 2 (Real) (N=12)
Skin surgery (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Routine skin surgery for the past 30 years
Transient ischemic attack-like symptoms (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real Then Sham - Month 1 (Real) (N=13) | Sham Then Real - Month 1 (Sham) (N=12) | Real Then Sham - Month 2 (Sham) (N=13) | Sham Then Real - Month 2 (Real) (N=12)
Temporary feeling of numbness or worsening in sensory scores (General disorders) | 3 (6) | 3 (22) | 2 (3) | 5 (10)
Temporary reduction in grip strength (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Temporary increase in Modified Ashworth scale scores (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Temporary increase in pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Temporary skin irritation (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (3) | 2 (4) | 1 (1)
Temporary swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Other (General disorders) | 2 (3) | 0 (0) | 2 (2) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT03318341/Prot_SAP_000.pdf